CLINICAL TRIAL: NCT07396363
Title: The Effect of Psychoeducational Psychotherapy on Neurocognitive Functions, Quality of Life, And Emotion Regulation in Adolescents Diagnosed With Bipolar Disorder: A Randomized Controlled Trial
Brief Title: Psychoeducational Psychotherapy in Adolescent Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ezgi Karagoz Tanigor M.D., Doctor in Child and Adolescent Psychiatry department, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 354-SBKAEK
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Disorder (BD)
Keywords: Bipolar Disorder; emotion regulation; neurocognition; quality of life; irritability
MeSH Terms: conditions — Bipolar Disorder; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducational psychotherapy (PEP) (Experimental): PEP is a structured, manualized, family-focused psychotherapy based on cognitive behavioral therapy (CBT). Participants were invited to participate in weekly parent and child sessions over a 12-week period. Each session lasted approximately 45-50 minutes, with a total of 24 sessions available throughout the trial. Parental involvement was incorporated into every PEP session, with parents joining for 5-10 minutes at the beginning of each child session to discuss the child's progress and for another 5-10 minutes at the end to review newly introduced material.
  Interventions: Behavioral: Psychoeducational psychotherapy (PEP)
- Control (No Intervention): Control group who received routine treatment and care.

INTERVENTIONS:
Behavioral: Psychoeducational psychotherapy (PEP) — PEP is a structured, manualized, family-focused psychotherapy based on cognitive behavioral therapy (CBT). Participants were invited to participate in weekly parent and child sessions over a 12-week period. Each session lasted approximately 45-50 minutes, with a total of 24 sessions available throughout the trial. Parental involvement was incorporated into every PEP session, with parents joining for 5-10 minutes at the beginning of each child session to discuss the child's progress and for another 5-10 minutes at the end to review newly introduced material.
  Arms: Psychoeducational psychotherapy (PEP)

SUMMARY:
This study evaluated the effects of psychoeducational psychotherapy (PEP) on neurocognitive functions, symptomatology, quality of life, and emotion regulation in euthymic adolescents with bipolar disorder (BD). Thirty-two adolescents with BD were randomized, with 16 receiving PEP. Assessments included the Wisconsin Card Sorting Test, Stroop Test, Pediatric Quality-of-Life Inventory, Difficulties in Emotion Regulation Scale (DERS), Affective Reactivity Index, Young Mania Rating Scale, and Children's Depression Rating Scale.

DETAILED DESCRIPTION:
This study aimed to examine the impact of PEP on neurocognitive performance, symptom levels, quality of life, and emotion regulation among euthymic adolescents diagnosed with BD. A total of 32 adolescents meeting diagnostic criteria for BD were randomly assigned to either an intervention group (n = 16), which received PEP, or a control group receiving standard care. Participants were evaluated using a comprehensive assessment battery that included the Wisconsin Card Sorting Test and the Stroop Test to measure executive functioning; the Pediatric Quality-of-Life Inventory to assess well-being; the DERS and the Affective Reactivity Index for emotional functioning; and the Young Mania Rating Scale and Children's Depression Rating Scale to evaluate mood symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 12 and 18 years who were diagnosed with BD (Bipolar Disorder)

Exclusion Criteria:

* Presence of chronic medical disorders, a clinical diagnosis of autism spectrum disorder, mental retardation or intellectual disability (according to developmental/academic history and clinical examination), past or current epilepsy, brain injury, and cerebral palsy

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
the Difficulties in Emotion Regulation Scale (DERS) | 12 weeks
  The Difficulties in Emotion Regulation Scale (DERS) assesses emotion regulation (ER) problems in adolescents across six domains: goals, strategies, impulsivity, awareness, clarity, and non-acceptance. Higher scores reflect greater ER difficulties. The Turkish version demonstrated good reliability and validity.

SECONDARY OUTCOMES:
Wisconsin Card Sorting Test | 12 weeks
  WCST is a test reflecting set-shifting which is defined as the flexibility in responses due to changes in reinforcement
The Pediatric Quality of life Inventory (PedsQL) | 12 weeks
  The PedsQL scale was used to assess problems within the multidimensional health-related quality of life in the last month. This is a modular instrument that is designed to measure health-related quality of life (HRQOL) among children and adolescents aged 2 to 18 years
Affective Reactivity Index-Child and Parent Forms | 12 weeks
  The Affective Reactivity Index-Child and Parent Forms is a scale developed for the evaluation and monitoring of irritability according to the reports of children and parents. Total scores range from 0 to 12, with higher scores indicating greater levels of irritability and thus a worse clinical outcome.
Young Mania Rating Scale | 12 weeks
  The Young Mania Rating Scale is an eleven item, likert-type scale that evaluates the symptoms of mania over the previous 48 hours or week, according to clinical observations and patient reports.The total score obtained from the scale ranges from 0 to 60, with higher scores indicating more severe manic symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Can not be shared due to ethical concerns

REFERENCES:
- [Result] Kowatch RA, Fristad M, Birmaher B, Wagner KD, Findling RL, Hellander M; Child Psychiatric Workgroup on Bipolar Disorder. Treatment guidelines for children and adolescents with bipolar disorder. J Am Acad Child Adolesc Psychiatry. 2005 Mar;44(3):213-35. doi: 10.1097/00004583-200503000-00006. PMID 15725966
- [Result] Bauer IE, Frazier TW, Meyer TD, Youngstrom E, Zunta-Soares GB, Soares JC. Affective Processing in Pediatric Bipolar Disorder and Offspring of Bipolar Parents. J Child Adolesc Psychopharmacol. 2015 Nov;25(9):684-90. doi: 10.1089/cap.2015.0076. Epub 2015 Oct 15. PMID 26468988